CLINICAL TRIAL: NCT00275574
Title: Acupuncture for the Treatment of Non-Cyclical Breast Pain
Brief Title: Acupuncture for Non-cyclical Breast Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Lori Thicke, APRN CNS, Mayo Clinic
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1975-02
Record Dates: First submitted 2006-01-10; First posted 2006-01-12 (Estimated); Last update posted 2016-01-01 (Estimated); Status verified 2015-12

CONDITIONS: Breast Pain
MeSH Terms: conditions — Mastodynia | interventions — Acupuncture Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- acupuncture (Experimental): four acupuncture treatments over a period of two weeks
  Interventions: Procedure: acupuncture

INTERVENTIONS:
Procedure: acupuncture — acupuncture

SUMMARY:
Breast pain or mastalgia is a common and troublesome symptom for many women. Whereas cyclical breast pain related to hormonal fluctuations can frequently be treated, non-cyclical breast pain can go untreated due to its various etiologies and non-specific presentation. Acupuncture is an ancient form of Chinese medicine that has been used for centuries to treat a vast array of illnesses and conditions. Research has shown that acupuncture has a link to a release of endorphins and other chemicals in the central nervous system. Thus, it is thought to help relieve pain. To date, there has been minimal research using acupuncture for breast pain. This pilot of 30 women will seek to determine whether four acupuncture treatments over a period of two weeks will significantly lower the level of pain experienced by these participants. Additionally, we will evaluate quality of life measures.

ELIGIBILITY:
* Female
* greater than 18 years
* non-cyclical unilateral or bilateral breast pain occurring daily, Greater than or equal to 2 on the BPI (average pain question)
* pain for more than 3 months
* satisfactory (non-suspicious for malignancy) breast examination within one year of enrollment (need documentation from physician or advanced practice nurse)
* satisfactory (non-suspicious for malignancy) mammogram and/or ultrasound within one year if Greater than 35 years(need written report to verify)
* able to return for acupuncture two times a week for two weeks
* speak and understand English
* hormone replacement therapy discontinued > 3 months

Ages: 18 Years to 100 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2003-04; Primary Completion 2009-08 (Actual); Study Completion 2009-08 (Actual)

PRIMARY OUTCOMES:
Four acupuncture treatments over a period of two weeks can improve non-cyclical breast pain | two weeks

CONTACTS AND LOCATIONS:
Overall Officials: Lori A. Thicke, R.N., M.S., Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States